CLINICAL TRIAL: NCT02135419
Title: ANCHOR Study: Anal Cancer/HSIL Outcomes Research Study
Brief Title: Treatment in Preventing Anal Cancer in Patients With HIV and Anal High-Grade Lesions
Acronym: ANCHOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); University of California, San Francisco (Other); University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMC-A01; NCI-2014-00636 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-A01 (Other: AIDS Malignancy Consortium); AMC-A01 (Other: CTEP); U01CA121947 (NIH); UM1CA121947 (NIH); ANCHOR (Other: AIDS Malignancy Consortium)
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Anal Cancer; High-grade Squamous Intraepithelial Lesion; HIV Infection; Human Papilloma Virus Infection
Keywords: anal cancer; high-grade squamous intraepithelial lesion; anal HSIL; HIV; HIV/AIDS; human papillomavirus; HPV
MeSH Terms: conditions — Anus Neoplasms; Squamous Intraepithelial Lesions; HIV Infections; Papillomavirus Infections; Acquired Immunodeficiency Syndrome | interventions — Imiquimod; Fluorouracil; Light Coagulation; Laser Therapy; Watchful Waiting; Observation

STUDY DESIGN:
Intervention Model Description: All participants are evaluated with high resolution anoscopy and anal cytology every 6 months during study participation. Participants randomized to treatment undergo biopsy of anal HSIL at each 6-month visit, and receive topical or ablative therapies for incident anal HSIL lesions. Active monitoring participants undergo close observation, with biopsy of anal HSIL at annual visits. Participants undergo biopsy of lesions at any time cancer is suspected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (treatment) (Experimental): Patients are directed to receive either topical or ablative treatment at the discretion of the clinician. Patients receiving topical treatment apply imiquimod intra-anally, peri-anally or both thrice weekly for up to 16 weeks, fluorouracil twice daily for 5 days every 2 weeks for up to 16 weeks, or trichloroacetic acid every 3 weeks up to 12 weeks. Patients receiving ablative treatment using infrared photocoagulation therapy, hyfrecation/electrocautery (thermal ablation therapy), or laser therapy. Patients may undergo excision under anesthesia if the clinician believes none of the other treatment approaches will be effective. The number and timing of such treatments will be at the discretion of the investigator. Patients with persistent HSIL should continue a protocol-approved treatment or a new protocol treatment should be considered. All participants will have samples collected for laboratory biomarker analysis.
  Interventions: Drug: imiquimod; Drug: fluorouracil; Device: infrared photocoagulation therapy; Device: thermal ablation therapy; Device: laser therapy; Other: clinical observation; Other: laboratory biomarker analysis
- Arm II (active monitoring) (closed since SEP2021) (Active Comparator): Patients undergo active monitoring with examinations for clinical observation every 6 months. Every 12 months, patients undergo biopsies of visible lesions. Patients have cytology sampling performed at every visit. All participants will have samples collected for laboratory biomarker analysis.
  Interventions: Other: clinical observation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imiquimod — Applied topically
  Other Names: Aldara; IMQ; R 837
  Arms: Arm I (treatment)
Drug: fluorouracil — Applied topically
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU; Efudex
  Arms: Arm I (treatment)
Device: infrared photocoagulation therapy — Undergo infrared coagulation
  Other Names: infrared coagulation; IRC
  Arms: Arm I (treatment)
Device: thermal ablation therapy — Undergo hyfrecation/electrocautery therapy
  Arms: Arm I (treatment)
Device: laser therapy — Undergo laser therapy
  Other Names: therapy, laser
  Arms: Arm I (treatment)
Other: clinical observation — Undergo active monitoring (High Resolution Anoscopy [HRA]) with biopsies
  Other Names: observation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The randomized phase of the trial compared topical or ablative treatment with active monitoring in preventing anal cancer in patients with human immunodeficiency virus (HIV) and high-grade squamous intraepithelial lesions (HSIL). Anal HSIL is tissue in the anal canal that has been damaged by infection with human papillomavirus (HPV) and is at risk for turning into anal cancer.

The ANCHOR Data Safety Monitoring Board (DSMB) determined that the primary study endpoint was completed, based on the data and statistical analysis presented to them on 07SEP2021.

In the post-randomization phase of this trial, all enrolled participants are offered treatment for HSIL and/or follow-up, at the participant's choice.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: The primary objective of this study has been completed for efficacy.

I. To determine the effectiveness of treating anal HSIL to reduce the incidence of anal cancer in human immunodeficiency virus (HIV)-infected men and women.

SECONDARY OBJECTIVES:

I. To determine the safety of infrared coagulation (IRC), electrocautery, imiquimod, laser and 5- fluorouracil treatments for anal HSIL.

II. To assess the responsiveness (sensitivity to change) and clinical significance of the ANCHOR Health-Related Symptom Index (A-HRSI) subscales by comparing change scores within groups of participants as defined by participant responses to the participant global impression of change (PGIC) item. (completed FEB2020)

TERTIARY OBJECTIVES:

Collect clinical specimens and data to create a bank of well-annotated specimens that will enable correlative science:

I. Identification of viral factors in HSIL progression to cancer; II. Identification of host factors in HSIL progression to cancer; III. Identify host and viral biomarkers of progression from HSIL to cancer; IV. Identify medical history and behavioral risk factors for HSIL progression to cancer.

QUALITY OF LIFE OBJECTIVES (completed FEB2022) I. Primary QOL Objective: To compare arms in terms of changes in physical symptoms and impacts from T2 to T3, adjusting for T1.

ANCILLARY (COVID SUPPLEMENT) SUBSTUDY OBJECTIVES:

I. Determine the prevalence of SARS-CoV-2 detection in anal and oropharyngeal swabs among people living with HIV (PLWH) being screened for and enrolled in the ANCHOR study.

II. Determine the relationship between prevalent anal SARS-CoV-2 positivity, anal HPV infection, and anal high-grade squamous intraepithelial lesions (HSIL).

III. Determine the 6-month incidence of SARS-CoV-2 detection in anal and oropharyngeal swabs among participants in the active monitoring arm being assessed for the first time for treatment and individuals already enrolled in the COVID substudy under protocol version 15.0.

IV. Determine the relationship between prevalent or incident SARS-CoV-2 detection and regression of anal HPV infection or HSIL among active monitoring arm participants already enrolled in the COVID substudy under protocol version 15.0, and those who continue the protocol and who choose not to be treated at visit 101.

OUTLINE: The randomized strategy to study the efficacy of HSIL treatment to reduce the risk of progression to anal cancer, as compared to active monitoring, was discontinued for all participants.

Patients are randomized to 1 of 2 treatment arms. (accrual closed SEP2021)

ARM I: Patients are directed to receive either topical or ablative treatment at the discretion of the clinician. Patients receiving topical treatment apply topical imiquimod intra-anally, peri-anally or both thrice weekly for up to 16 weeks, or topical 5-fluorouracil twice daily for 5 days every 2 weeks for up to 16 weeks. Patients receiving ablative treatment using infrared coagulation, hyfrecation/electrocautery, or laser. Patients may undergo excision under anesthesia if the clinician believes none of the other treatment approaches will be effective. The number and timing of such treatments will be at the discretion of the investigator. Patients with persistent HSIL should continue a protocol-approved treatment or a new protocol treatment should be considered.

ARM II: Patients undergo active monitoring with HRA examinations and anal cytology every 6 months. Every 12 months, patients undergo biopsies of visible lesions.

Participants on both arms are to be followed for up to 5 years after randomization of the last participant.

Post-randomization phase: Individuals in the treatment arm may continue treatment, and participants in the active monitoring arm are offered treatment. If upon assessment participants continue to have HSIL but do not intend to get treatment, they will be monitored for the potential for disease progression to anal cancer.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive. Documentation of HIV-1 infection by means of any one of the following: 1) Documentation of HIV diagnosis in the medical record by a licensed health care provider; 2) Documentation of receipt of ART by a licensed health care provider (receipt of at least two agents is required); 3) HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL; or, 4) Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay.
* Biopsy-proven HSIL at baseline
* At least one focus of HSIL must be identified that is not within a condyloma that may be treated after enrollment into the study
* For females, documentation that the participant is being followed for cervical cytology (if having a cervix) and/or HPV testing per current ASCCP guidelines, and visual examination of the vulva, vagina, and cervix to rule out cancer/suspicion for cancer within 12 months prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1 (Karnofsky >= 70%)
* Life expectancy of greater than 5 years
* Absolute neutrophil count: >= 750/mm^3
* Platelets: >= 75,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Women of childbearing potential must have a negative urine pregnancy test within 7 days of initiating study treatment if they have been randomized to the treatment arm; all women of childbearing potential must agree to use a reliable birth control method (oral contraceptive pills, intrauterine device, Nexplanon, DepoProvera, or permanent sterilization, etc., or another acceptable method as determined by the investigator) during the entire period of the trial (5 years or more), and must not intend to become pregnant during study participation and for 3 months after treatment is discontinued; all participants must be willing to comply with an acceptable birth control regimen as determined by the Investigator
* Men randomized to the treatment arm should not father a baby while receiving topical treatment during this study. Men who could father a child must agree to use at least one form of birth control during or continued abstinence from heterosexual intercourse if receiving topical treatment during the study, and for 2 weeks after stopping topical treatment.
* Ability to understand and the willingness to sign a written informed consent document
* Participant is willing to be randomized and able to comply with the protocol
* Clinician is comfortable with either following patient for up to 5 years without therapy or treating patient for up to 5 years

Exclusion Criteria:

* Inability to provide informed consent
* Patients who are receiving any other immunomodulatory investigational agents (replacement doses of steroids for adrenal insufficiency or treatment with prednisone ≤5 mg/day is permitted) within the 4 weeks before randomization enrollment, other than investigational antiretroviral agents for HIV, or investigational or approved agents for Hepatitis C.
* History of anal cancer, penile, vulvar, vaginal or cervical cancer, or signs of these cancers at baseline.
* Treatment or removal of HSIL less than 6 months prior to randomization.
* Participant has symptoms related to HSIL and would benefit more from immediate treatment than from entry into the study and potential for randomization to active monitoring arm
* Current systemic chemotherapy or radiation therapy that potentially causes bone marrow suppression that would preclude safe treatment of HSIL
* Participants who only have a single HSIL lesion that is likely to be removed entirely with the initial screening biopsy
* Warts so extensive that they preclude the clinician from determining the extent and location of HSIL
* Participant plans to relocate away from the study site to a location without an ANCHOR study site during study participation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4446 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — AIDS Malignancy Consortium
Locations (25):
- United States (24):
  - UCLA CARE Clinic, Los Angeles, California
  - UCLA School of Nursing, Los Angeles, California
  - DAP Health, Palm Springs, California
  - University of California at San Francisco Anal Dysplasia Clinic, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Public Health, Denver, Colorado
  - Capital Digestive Care, Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - ACC Clinic, Jackson Hospital, Miami, Florida
  - University of Miami Miller School of Medicine - Sylvester Cancer Center, Miami, Florida
  - Grady Health System, Atlanta, Georgia
  - Anal Dysplasia Clinic MidWest, Chicago, Illinois
  - University Medical Center New Orleans, New Orleans, Louisiana
  - CrescentCare Health, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Fenway Health, Boston, Massachusetts
  - Rutgers University New Jersey Medical School, Newark, New Jersey
  - Cornell Clinical Trials Unit, Chelsea Center, New York, New York
  - Laser Surgery Care, New York, New York
  - Montefiore - Albert Einstein College of Medicine, The Bronx, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - The Polyclinic, Seattle, Washington
- University of Puerto Rico, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
A CDISC-mapped, de-identified version of the study data with appropriate documentation (data dictionary, annotated static copies of electronic case report forms, clinical protocol, informed consent document) of the data elements will be made available via a public data repository: the AIDS Malignancy Consortium (AMC) Data Commons.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will only be shared with external investigators following conclusion of all participant data collection and the acceptance of a manuscript(s) that addresses all trial objectives, via release of the data to a public data repository, anticipated to occur on or after August 2025. Data will be available according to the archival terms of the AMC Data Commons.
Access Criteria: Qualified researchers with plans approved by the AMC Executive Committee who have entered into a Data Use Agreement (DUA) with the AMC will be granted data access. Research plans may include, but are not limited to, research on HIV/AIDS, anal HSIL screening and/or treatment, HPV-associated malignancies, anal cancer, and associated conditions.

REFERENCES:
- [Background] Lee JY, Lensing SY, Berry-Lawhorn JM, Jay N, Darragh TM, Goldstone SE, Wilkin TJ, Stier EA, Einstein M, Pugliese JC, Palefsky JM; ANCHOR Investigators. Design of the ANal Cancer/HSIL Outcomes Research study (ANCHOR study): A randomized study to prevent anal cancer among persons living with HIV. Contemp Clin Trials. 2022 Feb;113:106679. doi: 10.1016/j.cct.2022.106679. Epub 2022 Jan 10. PMID 35017115
- [Result] Palefsky JM, Lee JY, Jay N, Goldstone SE, Darragh TM, Dunlevy HA, Rosa-Cunha I, Arons A, Pugliese JC, Vena D, Sparano JA, Wilkin TJ, Bucher G, Stier EA, Tirado Gomez M, Flowers L, Barroso LF, Mitsuyasu RT, Lensing SY, Logan J, Aboulafia DM, Schouten JT, de la Ossa J, Levine R, Korman JD, Hagensee M, Atkinson TM, Einstein MH, Cracchiolo BM, Wiley D, Ellsworth GB, Brickman C, Berry-Lawhorn JM; ANCHOR Investigators Group. Treatment of Anal High-Grade Squamous Intraepithelial Lesions to Prevent Anal Cancer. N Engl J Med. 2022 Jun 16;386(24):2273-2282. doi: 10.1056/NEJMoa2201048. PMID 35704479
- [Derived] Barroso LF, Stier EA, Hillman R, Palefsky J. Anal Cancer Screening and Prevention: Summary of Evidence Reviewed for the 2021 Centers for Disease Control and Prevention Sexually Transmitted Infection Guidelines. Clin Infect Dis. 2022 Apr 13;74(Suppl_2):S179-S192. doi: 10.1093/cid/ciac044. PMID 35416975
- [Derived] Higashi RT, Rodriguez SA, Betts AC, Tiro JA, Luque AE, Rivera R, Barnes A. Anal cancer screening among women with HIV: provider experiences and system-level challenges. AIDS Care. 2022 Feb;34(2):220-226. doi: 10.1080/09540121.2021.1883512. Epub 2021 Feb 17. PMID 33594934

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021)
Started | 2227 | 2219
Completed | 2071 | 2080
Not Completed | 156 | 139

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received assigned intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021) | Total
Number analyzed (Participants) | 2227 | 2219 | 4446
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (8.9) | 50.9 (9.0) | 50.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 342 | 354 | 696
  Male | 1885 | 1865 | 3750
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 594 | 502 | 1096
  Not Hispanic or Latino | 1582 | 1665 | 3247
  Unknown or Not Reported | 51 | 52 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 14 | 25
  Asian | 27 | 26 | 53
  Native Hawaiian or Other Pacific Islander | 4 | 8 | 12
  Black or African American | 935 | 939 | 1874
  White | 1017 | 1016 | 2033
  More than one race | 89 | 98 | 187
  Unknown or Not Reported | 144 | 118 | 262
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 110 | 110 | 220
  United States | 2117 | 2109 | 4226
CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — Absolute CD4 count at baseline
  cells/mm^3 | 602 [398 to 827] | 607 [410 to 837] | 604 [400 to 834]

OUTCOME MEASURES:

1. Primary Outcome: Anal Cancer Incidence
Description: Anal cancer incidence is calculated as the number of anal cancer cases detected per 100,000 person years
Time Frame: Time from randomization to diagnosis of anal cancer, assessed up to 5 years post randomization
Population: Participants who were randomized and received the assigned intervention
Measure: Number (95% Confidence Interval); unit: cases per 100,000 person years
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021)
Number analyzed (Participants) | 2227 | 2219
cases per 100,000 person years | 173 [90 to 332] | 402 [262 to 616]

2. Secondary Outcome: Incidence of Adverse Events for Each Treatment
Description: Participants who had at least one adverse event (serious or non-serious)
Time Frame: Up to 5 years after randomization
Population: Participants who received assigned intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021)
Number analyzed (Participants) | 2227 | 2219
Participants | 416 | 429

3. Secondary Outcome: Change in Physical Symptom Score From Baseline (2-7 Days Post Randomization) Until 4 Weeks Post Randomization
Description: The physical symptom score is made up of the sum of responses to whether or not the participant had any of the 9 physical symptoms: anal pain, pain other than anal pain, pain during bowel movements, constipation, bleeding from anus, itching in/around the anus, discharge (wetness) in anal area, burning sensations in the anal area, and urgency for bowel movements. Responses are 0- not at all, 1-a little bit, 2-somewhat, 3-quite a bit, 4-very much. Thus physical symptom score ranges from 0 to 36.
Time Frame: 4 weeks post randomization
Population: Participants who were randomized on the ANCHOR study and for whom physical symptom scores were obtained at baseline and 4 weeks post-randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021)
Number analyzed (Participants) | 46 | 38
score on a scale | -2.22 (4.69) | -0.08 (3.31)

4. Other Pre Specified Outcome: Viral Factors in HSIL Progression to Cancer
Description: Descriptive statistics will be used to describe the integration locus of HPV In the invasive cancers and whether they differ from those of the overlying HSIL. Descriptive statistics will also be used to determine if the loci differ in HSIL that have progressed and concurrent HSIL biopsies that did not progress. In each case only tissues that contain HPV 16 will be analyzed.
Time Frame: Up to 5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-09

5. Other Pre Specified Outcome: Host Factors in HSIL Progression to Cancer
Description: Linear models will be fitted for each gene. Moderated t-statistics, fold-change and the associated p values will be calculated for each gene. Since thousands of genes will be tested, false discovery rate (FDR)-adjusted values will be calculated using the Benjamini-Hochberg method. FDR values indicate the expected fraction of falsely declared differentially expressed (DE) genes among the total set of declared DE genes, i.e. FDR = 0.15 would indicate that 15% of the declared DE genes were expected to be false due to experimental noise instead of actual differential expression.
Time Frame: Up to 5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-09

6. Other Pre Specified Outcome: Host and Viral Biomarkers of Progression From HSIL to Cancer
Description: Biomarkers that are correlated with progression from anal HSIL to anal cancer
Time Frame: Up to 5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-09

7. Other Pre Specified Outcome: Behavioral Risk Factors for HSIL Progression to Cancer
Description: For each risk factor of interest, Fisher's exact test or Pearson's chi-square test will be used to determine if there is an association. Factors associated with invasive anal cancer at the 0.10 significance level will be incorporated into a logistic regression model to determine if they are independently associated with invasive anal cancer. Cox regression analyses will also be used to evaluate the association between risk factors and time to diagnosis of invasive anal cancer.
Time Frame: Up to 5 years after randomization
Reporting Status: Not Posted, anticipated posting 2026-09

8. Other Pre Specified Outcome: ANCHOR Study Health-Related Symptom Index (A-HRSI) Scale Responsiveness (Sensitivity to Change)
Description: Participants at follow-up timepoints were categorized into two sets of three groups based on PGIC and ECOG PS responses ("worse," "no change," "better"), with the primary responsiveness analysis using these three groups in a one-way analysis of variance (ANOVA).
Time Frame: A-HRSI and self-reported Patient Global Impression of Change (PGIC) scale and ECOG Performance Status (ECOG PS) item were administered at time of enrollment (T1) up until time of trial randomization (T2), and 71-112 days post-randomization (T3).
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Quality of Life Assessment Measured by the A-HRSI (Validated Tool)
Description: A-HRSI physical symptoms and physical impacts subscale change scores (T3 minus T2) using an analysis of covariance adjusting for the covariate baseline (T1) subscale to test for differences between arms at a one-sided 0.025 significance level with approximately 90% power.
Time Frame: A-HRSI completion occurred at 3 time points: Pre-randomization (T1), within 2-7 days (T2) and at 4 weeks of treatment/randomization (T3).
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization until up to 5 years after randomization
Arm/Group | Arm I (Treatment) | Arm II (Active Monitoring) (Closed Since SEP2021)
All-Cause Mortality (participants affected / at risk) | 55/2227 | 48/2219
Serious Adverse Events (participants affected / at risk) | 370/2227 | 375/2219
Other Adverse Events (participants affected / at risk) | 82/2227 | 60/2219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Treatment) (N=2227) | Arm II (Active Monitoring) (Closed Since SEP2021) (N=2219)
Lung Infection (Infections and infestations) | 31 | 27
Infections and Infestations, other (Infections and infestations) | 27 | 31
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 56 | 56
Myocardial Infarction (Cardiac disorders) | 15 | 11
Chest pain - cardiac (Cardiac disorders) | 9 | 4
Heart Failure (Cardiac disorders) | 5 | 10
Sepsis (Infections and infestations) | 18 | 10
Skin Infection (Infections and infestations) | 20 | 17
Urinary tract infection (Infections and infestations) | 11 | 4
Fracture (Injury, poisoning and procedural complications) | 13 | 5
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 17
Depression (Psychiatric disorders) | 7 | 6
Suicide attempt (Psychiatric disorders) | 4 | 5
Acute kidney injury (Renal and urinary disorders) | 4 | 9
Chronic kidney disease (Renal and urinary disorders) | 5 | 6
Anemia (Blood and lymphatic system disorders) | 4 | 3
Cardiac arrest (Cardiac disorders) | 1 | 7
Cardiac disorders - other (Cardiac disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 3 | 6
enterocolitis (Gastrointestinal disorders) | 1 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 7
Death NOS (General disorders) | 13 | 10
Cholecystitis (Hepatobiliary disorders) | 5 | 6
Anorectal infecton (Infections and infestations) | 4 | 1
Appendicitis (Infections and infestations) | 4 | 2
Appendicitis perforated (Infections and infestations) | 3 | 2
Bone infection (Infections and infestations) | 6 | 6
Bronchial infection (Infections and infestations) | 3 | 2
Enterocolitis infection (Infections and infestations) | 4 | 5
Soft Tissue Infection (Infections and infestations) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 4
Stroke (Nervous system disorders) | 11 | 14
Seizure (Nervous system disorders) | 1 | 5
Psychiatric disorders, other (Psychiatric disorders) | 4 | 2
Suicidal ideation (Psychiatric disorders) | 4 | 5
Supraventricular tachycardia (Cardiac disorders) | 1 | 4
Aortic valve disease (Cardiac disorders) | 1 | 3
Blood and lymphatic system disorders, other (Blood and lymphatic system disorders) | 1 | 2
Mitral valve disease (Cardiac disorders) | 1 | 2
Ventricular arrythmia (Cardiac disorders) | 0 | 2
Congenital, familial and genetic disorders, other (Congenital, familial and genetic disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Anal hemorrhage (Gastrointestinal disorders) | 1 | 1
Colonic Fistula (Gastrointestinal disorders) | 0 | 2
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 2
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Gastric hemorrhage (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastrointestinal disorder, other (Gastrointestinal disorders) | 0 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 2
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal infection (Gastrointestinal disorders) | 1 | 1
Device related infection (Infections and infestations) | 2 | 1
Joint infection (Infections and infestations) | 3 | 0
Meningitis (Infections and infestations) | 2 | 2
Pelvic infection (Infections and infestations) | 0 | 2
Shingles (Infections and infestations) | 0 | 3
Thrush (Infections and infestations) | 1 | 1
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Fever (General disorders) | 2 | 0
Flu-like symptoms (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 2 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 2
Hepatitis failure (Hepatobiliary disorders) | 1 | 2
Allergic reaction (Immune system disorders) | 1 | 1
Upper respiratory infection (Infections and infestations) | 7 | 2
Viremia (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Sudden death, NOS (General disorders) | 6 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Treatment) (N=2227) | Arm II (Active Monitoring) (Closed Since SEP2021) (N=2219)
Infections and Infestations, other (Infections and infestations) | 40 | 36
Cardiac Disorders, Other (Cardiac disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 2 | 2
Anal hemorrhage (Gastrointestinal disorders) | 4 | 1
Anal pain (Gastrointestinal disorders) | 19 | 3
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Gastrointestinal disorder, other (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Anorectal infection (Gastrointestinal disorders) | 2 | 2
Neoplasms, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Surgical and Medical procedures, other (Surgical and medical procedures) | 2 | 0
Hypertension (Vascular disorders) | 2 | 4
Anal fistula (Gastrointestinal disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Injury, poisoning and procedural complications, other (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive Disturbance (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Pregnancy, puerperium and perinatal conditions, other (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT02135419/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT02135419/ICF_001.pdf